CLINICAL TRIAL: NCT01461941
Title: A Phase 2 Study of E6005 in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E6005-J081-201
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
Keywords: Dermatitis; Atopic
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis | interventions — methyl 4-(((3-(6,7-dimethoxy-2-(methylamino)quinazolin-4-yl)phenyl)amino)carbonyl)benzoate

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Drug: 0.2% E6005 ointment (Experimental)
  Interventions: Drug: E6005
- Drug: 0.0% E6005 ointment (vehicle) (Placebo Comparator)
  Interventions: Drug: E6005 ointment (vehicle)

INTERVENTIONS:
Drug: E6005 — 0.0% E6005 ointment applied twice daily for 4 weeks (vehicle-controlled phase), and then, following 8-week is extension phase which all subjects receive 0.2% E6005 ointment twice daily. Subjects are randomized to either 0.2% E6005 ointment group or vehicle group at a ratio of 2:1.
  Arms: Drug: 0.2% E6005 ointment
Drug: E6005 ointment (vehicle) — 0.2% E6005 ointment applied twice daily for 4 weeks (vehicle-controlled phase), and then, following 8-week is extension phase which all subjects receive 0.2% E6005 ointment twice daily. Subjects are randomized to either 0.2% E6005 ointment group or vehicle group at a ratio of 2:1.
  Arms: Drug: 0.0% E6005 ointment (vehicle)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety profiles of E6005 ointment in patients with atopic dermatitis compared to vehicle. The pharmacokinetic profile after topical application of E6005 is also assessed.

ELIGIBILITY:
Inclusion Criteria

* Adults of both genders aged 20 to 64 years at the time when the written informed consent is obtained.
* Outpatients diagnosed with atopic dermatitis.

Exclusion Criteria

* Patients with a present illness of Kaposi's varicelliform eruption, scabies, molluscum contagiosum, impetigo contagious, psoriasis, connective tissue disorder, collagen disorder or Netherton's syndrome, etc., which could have an effect on the pathological evaluation of the atopic dermatitis.
* Patients with active infection that requires oral or intravenous administration of antibiotics, antifungal or antivirus agent/s at baseline.
* Patients with advanced disease or abnormal laboratory tests that would possibly affect the safety of the subject or the implementation of this study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Changes of pruritus score from baseline | From baseline through 12 weeks
Changes of eczema area and severity from baseline | From baseline through 12 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Nagoya, Aichi-ken
  - Urayasu-shi, Chiba
  - Fukuoka, Fukuoka
  - Asahikawa-shi, Hokkaido
  - Sapporo, Hokkaido
  - Yokohama, Kanagawa
  - Adachi-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Minato-ku, Tokyo
  - Shinagawa-ku, Tokyo